CLINICAL TRIAL: NCT05056610
Title: Bestimmung Des Einflusses Von Nahrungsmitteln Auf Die Darmschleimhaut Mit Der Konfokalen Laserendomikroskopie Und Humanen in Vitro Organoiden
Brief Title: Confocal Laser Endomicroscopy to Determine Influence of Food Antigens on Mucosal Integrity
Acronym: RDS_CLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, yurdagül zopf, Professor Dr., University of Erlangen-Nürnberg Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Friedrich-Alexander-University
Record Dates: First submitted 2021-07-26; First posted 2021-09-24 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Irritable Bowel Syndrome; Food Sensitivity; Healthy Controls
Keywords: confocal laser endomicroscopy; organoids; intestinal permeability
MeSH Terms: conditions — Irritable Bowel Syndrome; Food Intolerance

STUDY DESIGN:
Intervention Model Description: During confocal endomicroscopy food antigens are given on the duodenal mucosa. The response of the mucosa is evaluated by the entry of fluorescein into the intestinal lumen and cell shedding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with IBS or FI (Experimental): Food antigens are added to duodenal mucosa during CLE
  Interventions: Other: food antigens on duodenal mucosa
- healthy controls (Experimental): Food antigens are added to duodenal mucosa during CLE
  Interventions: Other: food antigens on duodenal mucosa

INTERVENTIONS:
Other: food antigens on duodenal mucosa — Administration of food antigens on duodenal mucosa and determining the response through confocal laser endomicroscopy

SUMMARY:
Irritable bowel syndrome (IBS) is mainly associated with food intolerance and presents a particular challenge in gastrointestinal practice. The clinical symptoms are often associated by patients with the consumption of certain foods. This leads to strict elimination diets, and often without identification of the triggering food. In particular, the avoidance of wheat yields a relief of the clinical symptoms in many patients. Nevertheless, it is unclear which components of wheat are responsible for the symptoms. Besides the glutens, other wheat proteins, such as the amylase trypsin inhibitors, but also carbohydrates are discussed as triggers of the diseases.

Confocal laser endomicroscopy (CLE) is a new diagnostic method for detecting the local effect of food on the mucosa. CLE enables microscopic assessment of the mucosa already during an endoscopic examination and also allows statements to be made about intestinal permeability through changes in the influx of fluorescein into the intestinal lumen. In the course of the study, diluted food solutions are applied to the mucosa after a detailed assessment of the mucosa via the endoscope. The changes in mucosa and permeability are observed and documented.

Tissue samples are then taken for histopathological assessment of the degree of inflammation. Further biopsies are taken and cultured in vitro to produce human organoids. The organoids are stimulated with the food. Changes in proliferation, gene and cytokine expression are determined.

The aim of the proposed project is to investigate the influence of the main allergens, e.g. wheat, soy, milk, yeast and chicken egg white on the intestinal mucosa. The data obtained will be compared with the histopathological findings and the in vitro data in the human organoid model.

The long-term goal is to establish a valid patient-based rapid detection method for the detection of the triggering substances in patients with IBS or food intolerances.

DETAILED DESCRIPTION:
Patients with IBS of unclear etiology, i.e. non-IgE mediated food intolerances (FI), often have a long course of suffering. It is not uncommon for patients to follow self-imposed strict diets to alleviate food-dependent intestinal and extraintestinal symptoms. However, these diets carry a high risk of malnutrition. In practice, an elimination diet followed by provocation of individual foods attempts to identify the triggers of the intolerances. However, since the reaction to the food antigens can occur with a delay and not infrequently a combination of several intolerances is present, the correct diagnosis is often difficult. This often leads to a massively reduced quality of life for the patients and repeated examinations, such as gastrointestinal endoscopies, which lead to the patient being hospitalised again.

In addition to medical approaches to alleviate the symptoms (drugs for diarrhoea, laxatives for constipation), an improvement is often achieved through a change in diet. Recently, there have been increasing reports that patients with IBS respond to a diet that is reduced in FODMAPs (fermentable oligo-, di- and monosaccharides as well as polyols) with a significant improvement in symptoms. Furthermore, patients with IBS often report significant symptom relief with adherence to a gluten-free diet (GFD), so that current estimates suggest that almost half of patients with IBS benefit from a GFD.

The introduction of CLE provides a new objective method for detecting changes at the cellular level.The CLE allows a microscopic assessment of the mucosa already during the endoscopic examination and thus enables an vivo histology, with an exact analysis of the intestinal mucosa.

Others already showed that stimulation of intestinal mucosa with food antigens causes an increased permeability and cell shedding in patients with FI (Fritscher-Ravens et al. Gastroenterology 2014). The response to food antigens can be visualized after administration of intravenous fluorescein and measurement of the release of fluroescein in the gut lumen. A major advantage of CLE is the direct local assessment of food antigens on the intestinal mucosa and the identification of patients who have a clinically relevant FI.

Hypothesis: We suggest that patients with IBS and/or FI react more strongly to mucosal applied food antigens than healthy controls due to an existing low-grade intestinal inflammation. We plan to apply wheat, soy, milk, yeast and chicken egg white during CLE and record cell shedding and fluorescein efflux in the gut lumen. Since many patients with IBS are known to respond positively to a wheat-free diet, we expect the strongest mucosal response especially after application of wheat.

The aim is to prove our hypothesis by the increased cell shedding and the increased efflux of fluorescein into the intestinal lumen.

After CLE, tissue samples are taken for routine histopathological analysis. In addition, mucosal biopsies are taken and used to isolate stem cells and generate in vitro organoids. These organoids are cultured and supplemented with food antigens and changes in proliferation, gene, cytokine and chemokine expression are determined.

The primary goal is

* the evaluation of CLE with histopathological data, this means the determination of patients who have a good match of histopathologically confirmed inflammation with the assessment of mucosal changes detrrmined in CLE
* to determine the number of patients with IBS who have an response or change in permeability after application of the food antigens (wheat, soy, milk, yeast, chicken egg white) in CLE

Secondary objectives are

* the identification of molecular parameters after stimulation of in vitro organoids with food antigens
* the correlation of data derived from in vitro organoids with in vivo assessment during CLE

The study is planned for a period of 2 years. 40 patients aged 18 years and older with IBS who have a clinical need for oesophago-gastroduodenoscopy, e.g. to diagnose IBS or to exclude inflammatory bowel disease, gastritis, eosinophilic oesophagitis or coeliac disease, will be included in the study. Furthermore, 20 healthy control subjects who come for preventive medical checkup will be included.

Food antigens are applied during oesophago-gastroduodenoscopy, starting in the distal duodenum and proceeding sequentially to the proximal duodenum. The application of food antigens is randomised. The biopsies are taken after the application of the food antigens from the duodenal mucosa and used for histopathological analysis or in vitro generation of organoids.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* patients with IBS who fulfil the criteria according to Rome IV
* patients with suspected IBS who undergo gastroduodenoscopy for diagnosis of IBS
* healthy controls with no suspicion of food intolerance and/or presented for screening with an indication for oesophago-gastrodudodenoscopy (e.g. medical preventive examination, exclusion of H. pylori or gastritis)

Exclusion Criteria:

* lack of written consent
* patients with known allergy to fluorescein.
* Patients with carcinoma, liver disease, proven bacterial overgrowth
* Patients with diabetes mellitus
* Patients with severe cardiovascular disease or multiple concomitant drug therapy (beta-blockers)
* Patients with wheat allergy
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Correlation of the intestinal barriere defects determined by CLE with histopathological data | 2 years
  Correlation of the histopathologically confirmed inflammation and mucosal damage with in vivo data evaluated by CLE. In vivo damage will be reported and evaluated by efflux of fluorescein into the gut lumen and endothel cell shedding.
Determination of patients with IBS and response to food antigens | 2 years
  Determination of numbers of patients with IBS who show a response or change in permeability after application of the food antigens (wheat, soy, milk, yeast, chicken egg white) in CLE

SECONDARY OUTCOMES:
in vitro stimulation of intestinal organoids | 2 years
  RNA and protein analysis by RNA arrays, real-time PCR, Western blots, and enzyme linked immunoassays from organoids that are stimulated with food antigens.
correlation of data between organoids and CLE | 2 years
  Correlation of data derived from in vitro organoids with in vivo assessment during CLE

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine 1, Hector Center for Nutrition, Exercise and Sports, Friedrich-Alexander-University Erlangen-Nuremberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No